CLINICAL TRIAL: NCT06632691
Title: Virtual Reality Headset and Acceptability of Rectosigmoidoscopy in Ulcerative Colitis: a Randomised Controlled Trial
Acronym: VIRTU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD23_0096
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Haemorrhagic Rectocolitis
Keywords: Haemorrhagic rectocolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectosigmoidoscopy with virtual reality headset (Experimental)
  Interventions: Device: Virtual reality headset
- Rectosigmoidoscopy without a virtual reality headset (No Intervention)

INTERVENTIONS:
Device: Virtual reality headset — Use of a virtual reality headset during rectosigmoidoscopy
  Arms: Rectosigmoidoscopy with virtual reality headset

SUMMARY:
Haemorrhagic rectocolitis is an inflammatory bowel disease that continuously affects the rectum and colon, with lesions that extend variably from the rectum into the upstream colon. This disease requires repeated assessment of both clinical activity (transcribed by the clinical Mayo score) and endoscopic activity. ACCEPT study showed that the acceptability of rectosigmoidoscopy is low, and the main determinants of this low acceptability were pain and bloating (51%) and embarrassment during the examination (30%).

Virtual reality headsets has analgesic and anxiolytic properties, thanks to specially designed virtual environments that apply different principles such as medical hypnosis, music therapy and cardiac coherence to enhance therapeutic action.

The aim of our project is to study the benefit of medical hypnosis provided by the use of a virtual reality headset in terms of tolerance of lower digestive endoscopy in patients with ulcerative colitis.

DETAILED DESCRIPTION:
Haemorrhagic rectocolitis is an inflammatory bowel disease that continuously affects the rectum and colon, with lesions that extend variably from the rectum into the upstream colon.

This disease requires repeated assessment of both clinical activity (transcribed by the clinical Mayo score) and endoscopic activity. Assessment of mucosal healing is one of the therapeutic objectives defined in the STRIDE II consensus, and requires regular repeat endoscopic examinations in these patients.

The aim of the ACCEPT study, which involved administering a questionnaire to 916 patients with chronic inflammatory bowel disease, was to assess patients; acceptability and perceived usefulness of examinations designed to assess the activity of chronic inflammatory bowel disease. This study showed that the acceptability of rectosigmoidoscopy is low, and the main determinants of this low acceptability were pain and bloating (51%) and embarrassment during the examination (30%).

The dominant approaches to addressing this issue focus on replacing rectosigmoidoscopy with less invasive tools such as ultrasound and faecal calprotectin. However, rectosigmoidoscopy is still unavoidable, particularly for rectal forms (poor performance of ultrasound, low reliability of faecal calprotectin).

Virtual reality headsets are now part of our everyday lives. Developed as part of the neurosciences, they have applications in healthcare (pain care, dementia, post-traumatic stress disorder, etc.), occupational risk prevention and leisure (escape games, video games).

This device has analgesic and anxiolytic properties, thanks to specially designed virtual environments that apply different principles such as medical hypnosis, music therapy and cardiac coherence to enhance therapeutic action.

This approach has been evaluated in endoscopy, to improve the tolerance of colorectal cancer screening colonoscopies. A Chinese study (Liu et al, Clinical medicine 2022), which included 120 patients in a randomised trial comparing the virtual reality headset with a headset that was switched off, showed that the headset that was switched on made it possible to gain a median of 2 points on the pain scale, to reduce skin conductance (an indirect marker of nervousness) and to improve patient satisfaction. We hypothesise that the gain in SR would be the same, with an examination that is reputed to be less painful than colonoscopy without anaesthetic.

The aim of our project is to study the benefit of medical hypnosis provided by the use of a virtual reality headset in terms of tolerance of lower digestive endoscopy in patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over with UC in the active phase or in remission of their disease
* Patient who has already undergone rectosigmoidoscopy without general anaesthetic
* Patient requiring rectosigmoidoscopy (with colonoscope and air insufflation) as part of routine care
* Patient able to follow the Clinical Investigation protocol and having given written informed consent to participate
* Patient affiliated to the social security system or entitled beneficiary

Exclusion Criteria:

* Patients with Crohn disease or indeterminate colitis
* Patients hospitalised with severe acute colitis, as defined by the truelove criteria.
* Patients with a stoma in place or with a history of colorectal resection.
* Patients with a contraindication to the use of the virtual reality headset:

  * Psychotic patients or patients diagnosed with psychiatric disorders
  * Patients with uncontrolled epilepsy
  * Patients with visual problems (lack of binocular vision, blindness) and/or hearing problems (deafness) that prevent them from using virtual reality.
* Patients taking part in another clinical research protocol having an impact on the objectives of the clinical investigation
* Patients already randomized in the clinical investigation
* Pregnant, parturient or breast-feeding patients
* Patients under guardianship, curatorship or deprived of their liberty
* Patient under activated protection mandate or family habilitation
* Patients under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured on a visual analogue scale | Immediately after the examination.
  Pain intensity measured on a visual analogue scale (VAS) ranging from 0 (no pain) to 10 (maximum intolerable pain) immediately after the examination.

CONTACTS AND LOCATIONS:
Overall Officials: Morgane AMIL, Principal Investigator — Centre Hospitalier Départemental Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No